CLINICAL TRIAL: NCT04593212
Title: Improving the Assessment of Microcirculatory Dysfunction in Septic Shock Patients Using Optical Coherence Tomography Angiography at the Bedside
Brief Title: Assessment of Microcirculatory Dysfunction in Septic Shock Patients by OCTA
Acronym: SshOCTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital da Luz, Portugal (Other)
Responsible Party: Sponsor
Other Study IDs: id.215
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Septic Shock Survivors
  Interventions: Diagnostic Test: Optical Coherence Tomography Angiography
- Septic Shock Non-Survivors
  Interventions: Diagnostic Test: Optical Coherence Tomography Angiography

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography Angiography — Evaluation of microcirculatory dysfunction by assessment of retinal and choroidal microvasculature with optical coherence tomography angiography (OCTA)

SUMMARY:
Purpose and rationale: Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection. Sepsis and septic shock are major public health problems killing one in every three patients. Microcirculatory dysfunction is frequent in septic shock. The duration and severity of this dysfunction have a prognostic impact by being associated with organ failure and mortality. Our study purposes to demonstrate the feasibility of optical coherence tomography angiography (OCTA) to improve assessment of microcirculatory dysfunction by showing that retinal and choroidal microcirculatory changes with prognostic impact are present during septic shock.

Primary objective: To characterize the alterations of retinal and choroidal microcirculation in septic shock.

We will test the hypothesis that retinal and/or choroidal microcirculation shows dysfunctional changes (lower vascular density, lower percentage of perfused small vessel, lower blood flow index and higher vascular heterogeneity) in septic shock patients.

Secondary objective: To test the prognostic value of retinal and choroidal microcirculatory dysfunction in septic shock.

We will test the hypothesis that higher magnitude and persistence of retinal and/or choroidal microcirculatory dysfunction beyond the successful macro-hemodynamic resuscitation are independent predictors of organ failure and mortality in septic shock patients.

Study type: Two sequential observational studies.

Study design: A cross-sectional case-control study followed by a prospective cohort study with a 90-days longitudinal follow-up period.

Study population: 165 septic shock patients and 30 healthy controls.

Study duration: 90 days from enrolment to final follow-up assessment. One to two years of enrolment.

DETAILED DESCRIPTION:
Purpose and rationale: Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection. Sepsis and septic shock are major public health problems killing one in every three patients. Microcirculatory dysfunction is frequent in septic shock. The duration and severity of this dysfunction have a prognostic impact by being associated with organ failure and mortality. Our study purposes to demonstrate the feasibility of OCTA to improve assessment of microcirculatory dysfunction by showing that retinal and choroidal microcirculatory changes with prognostic impact are present during septic shock.

Primary objective (specific aim 1): To characterize the alterations of retinal and choroidal microcirculation in septic shock.

We will test the hypothesis that retinal and/or choroidal microcirculation shows dysfunctional changes (lower vascular density, lower percentage of perfused small vessel, lower blood flow index and higher vascular heterogeneity) in septic shock patients.

Secondary objective (specific aim 2): To test the prognostic value of retinal and choroidal microcirculatory dysfunction in septic shock.

We will test the hypothesis that higher magnitude and persistence of retinal and/or choroidal microcirculatory dysfunction beyond the successful macro-hemodynamic resuscitation are independent predictors of organ failure and mortality in septic shock patients.

Study type: Two sequential observational studies.

Study design: A cross-sectional case-control study followed by a prospective cohort study with a 90-days longitudinal follow-up period.

Study population: 165 septic shock patients and 30 healthy controls. Power and sample size calculations: Based on sublingual percentage of perfused small vessel (PPV) difference previously reported between septic shock patients and healthy controls (60% vs. 95%), we estimate that we will need to enrol 27 patients and 27 controls to demonstrate the same difference at the retina and choroid. To show a PPV difference between survivors and non-survivors (70% vs. 46%) in the septic shock group, also based on previous reports at the sublingual microcirculatory level, we estimate that we will need to enrol 150 septic shock patients. These calculations assumed an alpha level of 0.05 and a power of 80%. Our Department admits about 200 septic shock patients annually, so to account for drop-outs and limitations with enrolment (10-20% refusal to participate) we decided to increase our enrolment goal by 10% to 165 septic shock patients and 30 healthy controls.

Recruitment and inform consent: Recruitment will take place at the Intensive Care Medicine Department of Hospital da Luz Lisboa. Patients admitted to the Department with the diagnosis of septic shock will be screened for eligibility. If the patients are eligible to participate, they will be invited to enrol in the study by the principal investigator or other ICU medical team member. The study objectives and procedures will be explained to them. If the patient agrees to participate in the study, a written informed consent will be sign before enrolment. If the patient is unable to give informed consent to participate in the study, it will be asked to the reference next of kin using the same procedures as described before.

Study duration: 90 days from enrolment to final follow-up assessment. One to two years of enrolment.

Study procedures:

Baseline Assessment: After confirmation of eligibility and enrolment in the studies, demographic data (age, gender), type of admission (urgent/elective, medical/surgical/trauma), patient origin (emergency department, ward, operation room), source of infection (lung, urinary tract, intra-abdominal, skin and soft tissues, others), prognostic scores (APACHE II, SAPS II) and organic dysfunction scores (SOFA, quick SOFA) will be collected at baseline for septic shock patients.

Study Assessments:

OCTA: OCTA examination will be performed daily to septic shock patients from day 1 (less than 24 hours after diagnosis) until successful shock resolution (weaning from vasopressors) or until a maximum of 7 days. The healthy controls will be submitted to a single OCTA evaluation. We will use the Cirrus 6000® OCTA system (ZEISS, Germany) and the interpretation of OCTA images will be performed by two independent specialized ophthalmologists blinded to the clinical condition of patients. Images will be stored at the device working station.

Hemodynamic assessment: Every septic shock patient will have a central venous catheter and an arterial line in place according to the standard of care. Daily, during or within a maximum of 1 hour of OCTA examination, we will record the values of temperature, heart rate, mean arterial pressure, capillary refill time, central venous pressure, cardiac index, pH, PaCO2, PaO2, PvCO2, SaO2, SvO2, haemoglobin, serum lactate, fluid balance, oxygen delivery, oxygen consumption and oxygen extraction ratio.

Vasoactive and sedo-analgesic drugs: Daily we will record the vasoactive and sedo-analgesic drugs administered to septic shock patients and its total daily dose until complete weaning (defined as 24 hours free of vasopressors). Daily vasopressor score will also be calculated as suggested by Póvoa, P. et al.

Ventilatory and renal replacement therapy support: Daily we will record the type of ventilatory support (oxygen therapy, high flow oxygen therapy, non-invasive ventilation, invasive ventilation) and of renal replacement therapy (continuous, sustained low-efficiency, intermittent) used, if needed, until complete weaning.

Data analysis: In both studies, we will perform a descriptive statistical analysis of studied variables. Comparisons between healthy controls (single OCTA) and septic shock patients (first OCTA) to address endpoints related to specific aim 1 will be performed using t-Student test or Mann-Whitney test as appropriate. To address endpoints related to specific aim 2, we will compare survivors to non-survivors by doing a survival analysis using Kaplan-Meyer curves and Cox proportional hazards multivariable regression with microcirculatory measures as predictors. Additional comparisons will be performed using χ2 test, t-Student test, Mann-Whitney test and logistic regression as appropriate. We will assess confounding by adding significant variables in the regression models. We intend to perform a prespecified subgroup analysis of septic shock patients by serum lactate <4mmol/L vs. ≥4mmol/L and <2mmol/L vs. ≥2mmol/L. The correlation between retinal and choroidal microcirculation variables and macrohemodynamic variables will be assessed by the Spearman rank correlation coefficient. Area under Receiver Operating Characteristic curve of OCTA for prognostic outcomes will be calculated. A p-value < 0.05 will be considered statistically significant. Statistical analysis will be performed with STATA® 15 (StataCorp, Texas, USA).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years-old
* septic shock diagnosis (defined by the presence of sepsis according to Sepsis-3 definition plus a SOFA score ≥ 3 points at cardiovascular system despite adequate volume resuscitation) less than 24 hours before the first OCTA assessment

Exclusion Criteria:

* Inability or willingness to provide informed consent from the patient or next of kin
* Shock due to any other cause without septic shock
* Bilateral eye absence
* Previously known retinopathy
* Previous retinal surgery or photocoagulation
* Pregnant women
* Participants with psychiatry disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Source population:
  1. Cross-sectional case-control study: we intend to enrol 30 septic shock patients and 30 healthy controls.
  2. Prospective cohort study: we intend to enrol 165 septic shock patients (the first 30 patients will be the same from the cross-sectional case-control study).
  The enrolment will take place from patients admitted to the Intensive Care Medicine Department of Hospital da Luz Lisboa, from February 2021 to February 2022. The healthy controls will be enrolled from our hospital staff.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Perfused Small Vessel (PPV) | Daily assessment from day 0 to a maximum of 7 days
  The absolute number of completely perfused small vessels (diameter < 20μm) divided by the absolute number of small vessels (diameter < 20μm).
28-days All-Cause Mortality | 28-days after enrollment

SECONDARY OUTCOMES:
Perfused Small Vessel Density (PVD) | Daily assessment from day 0 to a maximum of 7 days
  The percentage area occupied by the small vessels (diameter <20μm)
Blood Flow Index (BFI) | Daily assessment from day 0 to a maximum of 7 days
  The average flow signal
Heterogeneity Index | Daily assessment from day 0 to a maximum of 7 days
  The difference between the highest and the lowest BFI divided by the mean BFI
ICU mortality | 90-days after enrollment
Hospital mortality | 90-days after enrollment
ICU length of stay | 90-days after enrollment
Hospital length of stay | 90-days after enrollment
Ventilator free-days | 90-days after enrollment
Vasopressor free-days | 90-days after enrollment
Renal replacement therapy free-days | 90-days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: André Alexandre, MD, Principal Investigator — 11170
Locations (1):
- Hospital da Luz Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Backer D, Cecconi M, Lipman J, Machado F, Myatra SN, Ostermann M, Perner A, Teboul JL, Vincent JL, Walley KR. Challenges in the management of septic shock: a narrative review. Intensive Care Med. 2019 Apr;45(4):420-433. doi: 10.1007/s00134-019-05544-x. Epub 2019 Feb 11. PMID 30741328
- [Background] Lipinska-Gediga M. Sepsis and septic shock-is a microcirculation a main player? Anaesthesiol Intensive Ther. 2016;48(4):261-265. doi: 10.5603/AIT.a2016.0037. Epub 2016 Sep 23. PMID 27660252
- [Background] Ince C. Hemodynamic coherence and the rationale for monitoring the microcirculation. Crit Care. 2015;19 Suppl 3(Suppl 3):S8. doi: 10.1186/cc14726. Epub 2015 Dec 18. PMID 26729241
- [Background] Ait-Oufella H, Bourcier S, Lehoux S, Guidet B. Microcirculatory disorders during septic shock. Curr Opin Crit Care. 2015 Aug;21(4):271-5. doi: 10.1097/MCC.0000000000000217. PMID 26103150
- [Background] Ince C. The rationale for microcirculatory guided fluid therapy. Curr Opin Crit Care. 2014 Jun;20(3):301-8. doi: 10.1097/MCC.0000000000000091. PMID 24758985
- [Background] De Backer D, Donadello K, Sakr Y, Ospina-Tascon G, Salgado D, Scolletta S, Vincent JL. Microcirculatory alterations in patients with severe sepsis: impact of time of assessment and relationship with outcome. Crit Care Med. 2013 Mar;41(3):791-9. doi: 10.1097/CCM.0b013e3182742e8b. PMID 23318492
- [Background] Spaide RF, Fujimoto JG, Waheed NK, Sadda SR, Staurenghi G. Optical coherence tomography angiography. Prog Retin Eye Res. 2018 May;64:1-55. doi: 10.1016/j.preteyeres.2017.11.003. Epub 2017 Dec 8. PMID 29229445
- [Background] Onishi AC, Fawzi AA. An overview of optical coherence tomography angiography and the posterior pole. Ther Adv Ophthalmol. 2019 Apr 3;11:2515841419840249. doi: 10.1177/2515841419840249. eCollection 2019 Jan-Dec. PMID 30984909
- [Background] Sambhav K, Grover S, Chalam KV. The application of optical coherence tomography angiography in retinal diseases. Surv Ophthalmol. 2017 Nov-Dec;62(6):838-866. doi: 10.1016/j.survophthal.2017.05.006. Epub 2017 Jun 1. PMID 28579550
- [Background] Alnawaiseh M, Ertmer C, Seidel L, Arnemann PH, Lahme L, Kampmeier TG, Rehberg SW, Heiduschka P, Eter N, Hessler M. Feasibility of optical coherence tomography angiography to assess changes in retinal microcirculation in ovine haemorrhagic shock. Crit Care. 2018 May 29;22(1):138. doi: 10.1186/s13054-018-2056-3. PMID 29843760
- [Background] Erikson K, Liisanantti JH, Hautala N, Koskenkari J, Kamakura R, Herzig KH, Syrjala H, Ala-Kokko TI. Retinal arterial blood flow and retinal changes in patients with sepsis: preliminary study using fluorescein angiography. Crit Care. 2017 Apr 10;21(1):86. doi: 10.1186/s13054-017-1676-3. PMID 28395665
- [Background] De Backer D, Creteur J, Preiser JC, Dubois MJ, Vincent JL. Microvascular blood flow is altered in patients with sepsis. Am J Respir Crit Care Med. 2002 Jul 1;166(1):98-104. doi: 10.1164/rccm.200109-016oc. PMID 12091178
- [Background] Sakr Y, Dubois MJ, De Backer D, Creteur J, Vincent JL. Persistent microcirculatory alterations are associated with organ failure and death in patients with septic shock. Crit Care Med. 2004 Sep;32(9):1825-31. doi: 10.1097/01.ccm.0000138558.16257.3f. PMID 15343008
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Povoa P, Salluh JI, Martinez ML, Guillamat-Prats R, Gallup D, Al-Khalidi HR, Thompson BT, Ranieri VM, Artigas A. Clinical impact of stress dose steroids in patients with septic shock: insights from the PROWESS-Shock trial. Crit Care. 2015 Apr 28;19(1):193. doi: 10.1186/s13054-015-0921-x. PMID 25928214